CLINICAL TRIAL: NCT03234764
Title: Longitudinal Follow-up Study for Food Allergies
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sharon Chinthrajah, Clinical Assistant Professor, Stanford University
Other Study IDs: 36616
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Food Allergy
Keywords: IgE; Allergy; Tolerance; Immunotherapy; Desensitization
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Sputum Buccal swab Saliva Urine Stool
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Immunotherapy

SUMMARY:
The purpose of this study is to evaluate the clinical usefulness of assessing specific human allergy antibodies and other immunologic parameters associated with the diagnosis, evolution, and management of allergic disease.

DETAILED DESCRIPTION:
The purpose of this study is to strengthen our ability to understand the long-term effects of food immunotherapy on the immune system and how it may induce tolerance to foods that participants were once allergic to. Investigators hope to determine tools and immunologic parameters that can help predict sustained desensitization and tolerance to food allergens following food immunotherapy. By evaluating the in-depth characteristics of allergy antibody populations and other immunologic parameters and comparing them to clinical disease, the investigators may uncover a more sound way to diagnose, follow and treat food allergic disease over time. Investigators will follow up with participants who underwent immunotherapy to food allergens as volunteers in clinical trials at the Sean N. Parker Center and assess whether they experience sustained desensitization to these foods in the long-term. Investigators will investigate the properties of the participants' immune cells and how they are affected over time by the ingestion of these food allergens. Investigators will follow the significance of different dosing regimens in terms of achieving tolerance. Differences in immune cell characteristics and other biological parameters may help predict the nature of a participant's tolerance to the food allergens and may help in the development of tools to determine permanent tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 6 months through 70 years who have previously undergone a food immunotherapy protocol only at our center.

Exclusion Criteria:

* None. However, if a participant becomes pregnant, their clinic visit may be postponed until after delivery and/or lactation period. These subject can postpone visits for one year and choose to skip visits during pregnancy and another year after (if breastfeeding).

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who underwent immunotherapy in clinical trial at the Sean N. Parker Center
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Immunological markers | February 2027
  IgE, IgG4, T cells

REFERENCES:
- [Background] Andorf S, Manohar M, Dominguez T, Block W, Tupa D, Kshirsagar RA, Sampath V, Chinthrajah RS, Nadeau KC. Observational long-term follow-up study of rapid food oral immunotherapy with omalizumab. Allergy Asthma Clin Immunol. 2017 Dec 21;13:51. doi: 10.1186/s13223-017-0223-8. eCollection 2017. PMID 29296107
- [Background] Andorf S, Manohar M, Dominguez T, Block W, Tupa D, Kshirsagar RA, Sampath V, Chinthrajah RS, Nadeau KC. Feasibility of sustained response through long-term dosing in food allergy immunotherapy. Allergy Asthma Clin Immunol. 2017 Dec 21;13:52. doi: 10.1186/s13223-017-0224-7. eCollection 2017. PMID 29296108